CLINICAL TRIAL: NCT03659929
Title: A Multicenter, Fixed-Dose, Double-Blind, Randomized Study to Evaluate the Efficacy and Safety of AR19 (Amphetamine Sulfate) in Adult Subjects (Ages 18-55) With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Adult Attention Deficit Hyperactivity Disorder (ADHD) Study With Amphetamine Sulfate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR19.004
Record Dates: First submitted 2018-08-29; First posted 2018-09-06 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Amphetamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: 20 mg/day (Experimental): Amphetamine Sulfate
  Interventions: Drug: Amphetamine Sulfate
- Arm 2: 40 mg/day (Experimental): Amphetamine Sulfate
  Interventions: Drug: Amphetamine Sulfate
- Arm 3: Placebo (Placebo Comparator): Placebo, no active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amphetamine Sulfate — active experimental AR19
  Other Names: AR19
  Arms: Arm 1: 20 mg/day; Arm 2: 40 mg/day
Drug: Placebo — Matching placebo
  Other Names: inactive drug
  Arms: Arm 3: Placebo

SUMMARY:
The purpose of the AR19.004 study is to assess the efficacy of AR19 compared to placebo using the Adult ADHD Investigator Symptom Rating Scale (AISRS)

DETAILED DESCRIPTION:
This is a randomized, fixed-dose, double-blind, multicenter trial to investigate the safety and efficacy of AR19 in the treatment of ADHD in adults from 18 through 55 years of age. Safety parameters and therapeutic effect will be evaluated throughout the trial. A target of 312 subjects is set for enrollment. Once subjects are determined to meet all inclusion criteria and were screened, they will be randomized to 20 or 40 mg AR19 daily or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female between 18 and 55 years of age, inclusive, at the time of Screening.
2. Meets criteria for diagnosis of ADHD using Conners' Adult ADHD Diagnostic Interview for Diagnostic and Statistical Manual of Mental Disorders (DSM-IV™) adapted for DSM-5™ (CAADID), including onset of ADHD symptoms before the age of 12.
3. Has an AISRS total score of ≥26 at Visit 2.
4. Has a clinician-administered Clinical Global Impression-Severity (CGI-S) score of 4 or greater at Visit 2.
5. In the clinical judgment of the Investigator, the subject needs pharmacological treatment for ADHD.
6. Must read and write English at a level sufficient to provide written informed consent and to complete study-related materials.
7. For subjects currently on a stable dose of allowed non-ADHD medication, there will be no expected changes in subject's medications during the study with the exception of medications listed in Section 5.9.2.
8. Males and females who are fertile and sexually active with a partner of the opposite sex must adhere to contraception requirements for the duration of the study as follows:

   * Females of childbearing potential must agree to be abstinent or to use highly effective forms of contraception.
   * Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months do not require contraception during the study.
   * Males , with female partners of childbearing potential must agree to be abstinent or use a medically acceptable form of contraception from screening through the end of study.

Exclusion Criteria:

1. Has a primary psychiatric diagnosis other than ADHD.
2. Has any other current secondary or co-morbid medical, psychiatric, or social condition which, in the opinion of the investigator, might compromise subject safety, or is likely to interfere with protocol compliance or to confound the assessment of safety or efficacy.
3. Has a history or current symptoms of bipolar disorder, schizophrenia, or psychotic disorder.
4. Has clinically significant cognitive impairment in the clinical judgment of the Investigator.
5. Has a Body Mass Index (BMI) of <17 or ≥39 kg/m2.
6. Has a Screening or Baseline triplicate-average blood pressure of ≥139 millimeter of mercury (mmHg) systolic or ≥89 mmHg diastolic. Blood pressure will be taken in triplicate, and the average will be used for evaluating entry criteria.
7. Is pregnant or breastfeeding, or is planning to become pregnant during the study.
8. Has a history of any of the following disorders:

   * Seizure disorder (excluding a history of isolated febrile seizures <6 years old),
   * Inadequately or not treated hypertension is defined as a subject who has blood pressure indicative of Stage 2 hypertension (systolic pressure ≥140 mmHg or diastolic pressure ≥90 mmHg). Subjects who are adequately treated must be on a stable dose of antihypertensive medications for 3 months prior to screening and their antihypertensive medications are not anticipated to change.
   * Untreated thyroid disease. Subjects with a history of thyroid disease who have been on a stable dose of thyroid hormone for at least three months are eligible to participate if their thyroid-stimulating hormone (TSH) does not fall in the excluded range, shown below in 14.
   * Glaucoma
   * Tourette's disorder, or chronic tics.
   * Subjects who have had gastrointestinal surgery or a procedure that involves:

     * Excision or partial excision of the esophagus, stomach, small and large intestine, liver, pancreas or biliary tree. Appendectomy, cholecystectomy and/or removal of gallstones in the bile ducts (as long as the ducts remain intact) are exceptions.
     * Reduction of the stomach volume without excision or partial excision of the stomach (e.g. restrictive surgery/procedure)
     * Obesity treatments that can affect gastrointestinal (GI) capacity or function, such as electrical stimulation systems, gastric balloon systems, and gastric external drainage systems
9. Has Electrocardiogram (ECG) or clinical evidence of the following:

   * Fridericia's corrected QT wave interval (QTcF) > 470 milliseconds (msec) for females, and > 450 msec for males
   * Atrial or ventricular hypertrophy
   * Intraventricular conduction defects other than incomplete right bundle branch block in the absence of other heart disease
   * Myocardial infarct, ischemia, or symptomatic coronary artery disease within 1 year prior to the Screening Visit
   * Clinically significant atrial or ventricular dysrhythmia; the heart must be in predominantly normal sinus rhythm
   * Second or third degree atrioventricular block
   * Heart failure
   * Functionally significant cardiac structural abnormality or valvular disease
   * Cardiomyopathy
   * Any other cardiovascular condition that the Investigator feels may predispose the subject to cardiovascular events (e.g. myocardial infarction, stroke) or arrhythmia
10. Known family history of sudden cardiac death in the absence of pre-existing heart disease.
11. Use of any psychotropic medication within 28 days of the Baseline visit except for ADHD medication. (Sedative hypnotics prescribed as a sleep aid at a stable dose for at least 28 days prior to Baseline, at bedtime only, are allowed during the study.)
12. Has used prohibited drugs or agents within 28 days of the Baseline visit through Study Visit 7. (Stimulant medications are allowed until 7 days before the Baseline visit.) Non-stimulant ADHD medications (guanfacine, bupropion, clonidine, and/or atomoxetine) are not allowed within 28 days of Visit 2 or at any time during the study. Note: Medications that are being taken for psychiatric or medical disorders other than ADHD should not be discontinued for the purpose of qualifying for study participation unless the medication is deemed medically unnecessary by the prescribing physician.
13. Has received an investigational drug within 60 days of the Screening visit.
14. Has an abnormal laboratory test value, vital sign, or other exam finding at Screening or Baseline that, in the opinion of the Investigator, warrants exclusion from the study. In addition, subjects with laboratory values listed below are considered exclusionary:

    * Serum aspartate transaminase (AST) or alanine transaminase (ALT) >1.5 × upper limit of normal (ULN)
    * Serum total bilirubin >1.5 × ULN unless due to Gilbert's Syndrome
    * Serum creatinine >1.3 × ULN
    * Glycosylated hemoglobin (HbA1c) ≥7.0%.
    * TSH <0.9 × lower limit of normal (LLN) or TSH >1.2 × ULN
15. Reports a history of hypersensitivity or intolerance to any formulation of amphetamine.
16. Reports a history of poor therapeutic response to any formulation of amphetamine or methylphenidate despite a clearly adequate trial (including dose and duration).
17. Is unable to swallow medication in capsule form.
18. Is unable or unwilling to follow directions of study staff or comply with all the testing and requirements of the protocol.
19. Has a positive urine drug result at Screening (with the exception of current ADHD stimulant therapy, if any). Note: subjects should be informed that they should not participate in the trial or submit to urine drug testing if they are using any controlled or recreational drug (other than a prescribed stimulant for ADHD), and non-use should be confirmed prior to testing.
20. Has a positive blood alcohol level at Screening. Note: subjects should be informed that alcohol consumed within 12 hours of screening may result in a positive test.
21. Has current or known history of drug or alcohol abuse within the past 12 months.
22. Has a history of human immunodeficiency virus (HIV), hepatitis B, or untreated hepatitis C infection. Note: subjects with a history of hepatitis C infection who have been treated and whose hepatitis C virus ribonucleic acid (HCV RNA) is currently undetectable are not excluded.
23. In the past 12 months, has had an intensity of suicidal ideation of greater than 1or any self-injurious behavior using the Columbia Suicide Severity Rating Scale at the Screening or Baseline visits.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Caras, MD, PhD, Study Director — Arbor Pharmaceuticals
Locations (31):
- United States (31):
  - 114: Pharmacology Research Institute, Encino, California
  - 133: Collaborative Neuroscience Network, Garden Grove, California
  - 124: Pharmacology Research Institute, Newport Beach, California
  - 121: CT Clinical Research Associates, Cromwell, Connecticut
  - 108: Meridien Research, Bradenton, Florida
  - 103: Gulfcoast Clinical Research Center, Fort Myers, Florida
  - 129: Sarkis Clinical Trials, Gainesville, Florida
  - 105: Meridien Research, Lakeland, Florida
  - 120: Meridien Research, Maitland, Florida
  - 130: Medical Research Group of Central Florida, Orange City, Florida
  - 123: APG Research, LLC, Orlando, Florida
  - 115: Clinical Neuroscience Solutions (CNS), Inc., Orlando, Florida
  - 104: Northwest Behavioral Research Center, Marietta, Georgia
  - 131: Advanced Clinical Research, Inc., Meridian, Idaho
  - 113: Capstone Clinical Research, Libertyville, Illinois
  - 134: Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - 128: Clinical Neurophysiology Services, Sterling, Michigan
  - 107: Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - 116: Alliance - Hassman Research Institute, Berlin, New Jersey
  - 127: Center for Emotional Fitness, Cherry Hill, New Jersey
  - 101: Princeton Medical Institute, Princeton, New Jersey
  - 118: Bioscience Research, LLC, Mount Kisco, New York
  - 119: Neurobehavioral Clinical Research, Inc., Canton, Ohio
  - 106: Summit Research Network, Portland, Oregon
  - 126: Coastal Carolina Research, Mt. Pleasant, South Carolina
  - 102: Clinical Neuroscience Solutions (CNS), Inc., Memphis, Tennessee
  - 132: Research Strategies of Memphis, Memphis, Tennessee
  - 125: Biobehavioral Research of Austin, Austin, Texas
  - 110: FutureSearch Trials of Dallas, Dallas, Texas
  - 117: Houston Clinical Trials, LLC, Houston, Texas
  - 109: Ericksen Research and Development, Clinton, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faraone SV, Childress A, Caras S, Arnold VK, Montano CB, Sarkis EH, Cutler AJ, Young JL. A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of AR19, a Manipulation-Resistant Formulation of Amphetamine Sulfate, in Adults With Attention-Deficit/Hyperactivity Disorder. J Clin Psychiatry. 2021 Aug 24;82(5):21m13927. doi: 10.4088/JCP.21m13927. PMID 34428356

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo, no active drug
  Placebo: Matching placebo
- Amphetamine Sulfate (20 mg/Day); Amphetamine Sulfate (40 mg/Day): Amphetamine Sulfate
  Amphetamine Sulfate: active experimental AR19
Period: Overall Study
Arm/Group | Placebo | Amphetamine Sulfate (20 mg/Day) | Amphetamine Sulfate (40 mg/Day)
Started | 106 | 107 | 107
Completed | 92 | 87 | 87
Not Completed | 14 | 20 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Amphetamine Sulfate (20 mg/Day) | Amphetamine Sulfate (40 mg/Day) | Total
Number analyzed (Participants) | 106 | 107 | 107 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (10.75) | 35.6 (10.28) | 33.5 (9.35) | 34.4 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 50 | 44 | 146
  Male | 54 | 57 | 63 | 174
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 13 | 14 | 41
  Not Hispanic or Latino | 92 | 94 | 93 | 279
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 6 | 1 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 13 | 13 | 15 | 41
  White | 80 | 89 | 88 | 257
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 4 | 1 | 11
ADHD Type [Count of Participants; unit: Participants]
  Inattentive | 14 | 19 | 20 | 53
  Hyperactive/Impulsive | 1 | 0 | 0 | 1
  Combined | 91 | 88 | 87 | 266

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Severity of Attention Deficit Hyperactivity (ADHD) Symptoms
Description: Change from baseline in severity of Attention Deficit Hyperactivity (ADHD) symptoms, as measured by the adult ADHD Investigator Symptom Rating Scale (AISRS), with a minimum score of 0, and maximum score of 54. Higher scores indicate more severe symptoms, or a worse outcome.
Time Frame: Week 5 (Visit 7)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Amphetamine Sulfate (20 mg/Day) | Amphetamine Sulfate (40 mg/Day)
Number analyzed (Participants) | 103 | 106 | 105
score on a scale | -11.1 (1.28) | -18.2 (1.28) | -18.1 (1.27)

2. Secondary Outcome: Change From Baseline to Visit 7 in AISRS Hyperactive and Inattentive Subscale Scores
Description: Items are scored as follows: 0 (none), 1 (mild), 2 (moderate), 3 (severe). The maximum total score for the scale is 54 points, with 27 points for each subscale (summed). The total score is the sum of the inattentive and hyperactive-impulsive subscales. Higher values represent more severe hyperactivity and/or inattentiveness.
Time Frame: Up to 5 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Amphetamine Sulfate (20 mg/Day) | Amphetamine Sulfate (40 mg/Day)
Number analyzed (Participants) | 103 | 106 | 105
score on a scale
  Hyperactivity/Impulsivity Subscale | -5.2 (0.61) | -8.3 (0.61) | -8.0 (0.6)
  Inattentive Subscale | -5.9 (0.74) | -9.9 (0.74) | -10.0 (0.74)

3. Secondary Outcome: Change in Clinical Global Impression of Severity (CGI-S) Score From Baseline
Description: CGI-Severity (CGI-S): The CGI-Severity (CGI-S) asks the clinician one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
Time Frame: Up to 5 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Amphetamine Sulfate (20 mg/Day) | Amphetamine Sulfate (40 mg/Day)
Number analyzed (Participants) | 103 | 106 | 105
score on a scale
  Visit 3 (Week 1) | -0.5 (0.1) | -0.9 (0.1) | -1.0 (0.1)
  Visit 4 (Week 2) | -0.7 (0.12) | -1.1 (0.12) | -1.3 (0.12)
  Visit 5 (Week 3) | -0.8 (0.12) | -1.4 (0.12) | -1.5 (0.12)
  Visit 6 (Week 4) | -0.8 (.12) | -1.4 (.12) | -1.5 (0.12)
  Visit 7 (End of Study/End of Treatment) | -0.9 (.13) | -1.5 (.13) | -1.5 (.13)

4. Secondary Outcome: Change in Clinical Global Impression of Improvement (CGI-I) Score From Baseline
Description: "Compared to the patient's condition at admission to the project [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment."
Time Frame: Up to 5 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Amphetamine Sulfate (20 mg/Day) | Amphetamine Sulfate (40 mg/Day)
Number analyzed (Participants) | 103 | 106 | 105
score on a scale
  Visit 3 (Week 1) | 3.3 (0.1) | 2.9 (0.1) | 2.8 (0.1)
  Visit 4 (Week 2) | 3.2 (0.11) | 2.6 (0.11) | 2.4 (0.11)
  Visit 5 (Week 3) | 3.0 (0.11) | 2.6 (0.11) | 2.4 (0.11)
  Visit 6 (Week 4) | 3.1 (0.11) | 2.5 (0.11) | 2.4 (0.11)
  Visit 7 (End of Study/End of Treatment) | 3.1 (0.12) | 2.5 (0.12) | 2.4 (0.12)

5. Secondary Outcome: Change in Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) Score From Baseline
Description: The Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) is a 75-item self-rating scale that assesses overall functioning (GEC) and 9 non-overlapping scales among 2 summary index scales (Metacognition Index [MI] and Behavioral Regulation Index [BRI]) that assess aspects of executive function and problems with self-regulation from the perspective of the individual.
  Subjects rate each item on a 3-point scale (1=Never, 2=Sometimes, or 3=Often) based on their experience in past month.
  The sum of 70 items yields the GEC raw score (range: 70-210), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥ 65 is considered abnormally elevated). The post-baseline GEC T-score is converted to a change from baseline T-score.
  A lower change from baseline GEC T-score (<0) represents a better outcome.
Time Frame: Up to 5 weeks
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo | Amphetamine Sulfate (20 mg/Day) | Amphetamine Sulfate (40 mg/Day)
Number analyzed (Participants) | 103 | 106 | 105
T-Score
  Global Executive Composite T-Score | -7.4 (1.33) | -13.6 (1.35) | -14.6 (1.31)
  Behavioral Regulation Index T-Score | -6.4 (1.15) | -11.5 (1.17) | -12.8 (1.14)
  Metacognition Index (MI) T-Score | -7.2 (1.32) | -13.4 (1.37) | -14.2 (1.33)
  Inhibit T-Score | -7.1 (1.22) | -11.3 (1.25) | -13.0 (1.21)
  Self-Monitor T-Score | -5.2 (1.10) | -10.6 (1.12) | -11.9 (1.09)
  Plan/Organize T-Score | -6.9 (1.30) | -12.2 (1.33) | -12.9 (1.29)
  Shift T-Score | -4.8 (1.13) | -9.8 (1.16) | -10.4 (1.13)
  Initiate T-Score | -5.0 (1.16) | -10.3 (1.19) | -11.2 (1.15)
  Task Monitor T-Score | -6.8 (1.33) | -12.6 (1.36) | -13.5 (1.32)
  Emotional Control T-Score | -3.9 (0.94) | -7.1 (0.96) | -8.0 (0.93)
  Working Memory T-Score | -7.5 (1.36) | -13.4 (1.40) | -14.8 (1.36)
  Organization of Materials T-Score | -4.3 (1.09) | -9.5 (1.12) | -10.0 (1.09)

ADVERSE EVENTS:
Time Frame: Collection of AE information started with the first dose of the study drug (Day 2) and continued through the post-withdrawal follow-up phone call (i.e., 7 days after Visit 7 [Week 5])
Arm/Group | Placebo | Amphetamine Sulfate (20 mg/Day) | Amphetamine Sulfate (40 mg/Day)
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/107 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/107 | 0/107
Other Adverse Events (participants affected / at risk) | 19/106 | 46/107 | 55/107
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=106) | Amphetamine Sulfate (20 mg/Day) (N=107) | Amphetamine Sulfate (40 mg/Day) (N=107)
Insomnia (Psychiatric disorders) | 4 | 9 | 10
Dry Mouth (Gastrointestinal disorders) | 4 | 6 | 12
Headache (Nervous system disorders) | 13 | 14 | 12
Nasopharyngitis (Infections and infestations) | 6 | 5 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 11 | 14
Palpitations (Cardiac disorders) | 2 | 2 | 7
Tachycardia (Cardiac disorders) | 0 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03659929/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT03659929/SAP_001.pdf